CLINICAL TRIAL: NCT02500251
Title: Belimumab-Based Plasma Cell Targeted Therapy to Impact Transplant Eligibility
Brief Title: Belimumab Impacting Transplant Eligibility
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: E. Steve Woodle (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, E. Steve Woodle, Director, Solid Organ Transplantation, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Belimumab
Record Dates: First submitted 2015-07-09; First posted 2015-07-16 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Renal Transplant Rejection
Keywords: Transplantation; belimumab; Velcade
MeSH Terms: interventions — belimumab; Bortezomib; Rituximab; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (5 subjects) (Experimental): Subjects will receive bortezomib and plasmapheresis.
  Interventions: Drug: Bortezomib; Drug: Plasmapheresis
- Group B (5 subjects) (Experimental): Subjects will receive belimumab, bortezomib, and plasmapheresis.
  Interventions: Drug: belimumab; Drug: Bortezomib; Drug: Plasmapheresis
- Group C (5 subjects) (Experimental): Subjects will receive belimumab, bortezomib, rituximab, and plasmapheresis.
  Interventions: Drug: belimumab; Drug: Bortezomib; Drug: Rituximab; Drug: Plasmapheresis

INTERVENTIONS:
Drug: belimumab — Belimumab will be administered per study protocol.
  Other Names: benlysta
  Arms: Group B (5 subjects); Group C (5 subjects)
Drug: Bortezomib — Bortezomib will be administered per study protocol.
  Other Names: Velcade
Drug: Rituximab — Rituximab will be administered per study protocol.
  Other Names: Rituxan
  Arms: Group C (5 subjects)
Drug: Plasmapheresis — Plasmapheresis will be administered per study protocol.

SUMMARY:
This study is a prospective, open label, phase I/II pilot study.

DETAILED DESCRIPTION:
This study is a prospective, open label, phase I/II pilot study. For Treatment Groups A and B, the duration of study will include a 5 month enrollment period and approximately 7 months of follow-up. For Treatment Group C, the duration of study will include a 3 month enrollment period and approximately 7 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 65 years of age, inclusive, with end-stage renal disease awaiting kidney transplantation.
2. Patient with eligible living donor will have: DSA against living donor of > 5,000 MFI or a positive T or B cell flow cytometry crossmatch.
3. Patient that is on the kidney transplant waiting list awaiting a deceased donor transplant and has an iAb of > 8,000 MFI or has a current or peak calculated panel reactive antibody (cPRA) >20%.
4. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
5. Female subject is either post-menopausal for one year prior to screening or surgically sterilized. Women of childbearing potential (WOCBP) must not become pregnant and so must be sexually inactive by abstinence (starting 2 weeks prior to the 1st belimumab and/or bortezomib dose) or use contraceptive methods with a failure rate of < 1% (starting 1 month prior to the 1st belimumab and/or bortezomib dose) for the duration of the study through 16 weeks after the last belimumab and/or bortezomib dose. WOCBP must have a negative urine or serum pregnancy test at screening and < 7 days prior to the first belimumab and/or bortezomib dose.
6. Male subjects, even if surgically sterilized (i.e., status post vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 16 weeks after the last dose of belimumab and/or bortezomib, or completely abstain from heterosexual intercourse.
7. Review of pre-transplant medical clearance by the patient's transplant nephrologist to assure the patient is medically acceptable for study entry.
8. Cardiac evaluation by transplant nephrologist with clearance documented in writing to participate in the study.

Exclusion Criteria:

1. Know hypersensitivity to bortezomib, boron or mannitol, rituximab, belimumab or any of its components.
2. Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
3. Subjects judged by the investigator to be at significant risk of failing to comply with the requirements of the protocol or unable to cooperate or communicate with the investigator.
4. Abnormal ECG with clinically significant ventricular arrhythmias or other conduction abnormality that in the opinion of the investigator warrants exclusion of the subject from the trial.
5. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (Appendix A), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any abnormality on ECG performed within 30 days of consent has to be documented by the investigator or the patient's transplant nephrologist as not medically relevant.
6. Patient has Grade 2 peripheral neuropathy by CTCAE criteria within 14 days before enrollment.
7. Patients with an absolute neutrophil count < 1,000/mm3 or platelet count < 75,000/mm3 within 30 days of consent.
8. Patient has received intravenous cyclophosphamide within 180 days prior to belimumab, any biologic investigational agent within 365 days prior to belimumab, or any non-biologic investigational agent within 30 days (or 5 half-lives, whichever is greater) prior to belimumab.
9. Receipt of a live vaccine within 30 days prior to initiation of study treatment.
10. Received blood transfusions within 30 days prior to trial entry.
11. Have any intercurrent significant medical (other than renal disease) or psychiatric illness that the investigator considers would make the candidate unsuitable for the study.
12. Have a historically positive HIV test or test positive for HIV within one year of consent.
13. Hepatitis status:

    a. Hepatitis B: Serologic evidence of current or past Hepatitis B (HB) infection based on the results of testing for HBsAg and anti-HBc as follows: i. Patients positive for HBsAg or HBcAb historically or on testing performed within one year of consent are excluded b. Hepatitis C: Positive test for Hepatitis C antibody with a detectable viral load on testing performed within one year of consent.
14. History of malignancy within the past 5 years that is not considered to be cured, with the exception of localized basal cell carcinoma of the skin (excised ≥ 2 years prior to randomization).
15. Evidence of severe liver disease with abnormal liver profile (aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin > 1.5 times upper limit of normal (ULN)) on testing performed within 30 days of consent.
16. Infection history: a)Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria). b) Hospitalization for treatment of infection within 60 days of Day 0. c) Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 0.
17. Pregnant or nursing (lactating) women and women who might become pregnant during the study.
18. Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.
19. Have a history of a primary immunodeficiency.
20. Have a significant IgG deficiency (IgG level < 400 mg/dl) or have an IgA deficiency (IgA level < 10 mg/dL).
21. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 0.
22. Have any other clinically significant abnormal laboratory value in the opinion of the investigator warrants exclusion of the subject from the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of belimumab as measured by percent reduction in iDSA and/or iAb | 7 months
  Maximal percent reduction in immunodominant DSA (iDSA) [highest titer DSA (MFI)] and/or immunodominant antibody (iAb) from pre-treatment to Day 151.

SECONDARY OUTCOMES:
Safety of belimumab as measured by toxicities and peripheral neuropathy | 7 months
  Overall safety of belimumab when used in the desensitization setting with bortezomib with or without rituximab (Incidence of grade 3 and above non-hematologic toxicities; Incidence of grade 4 hematologic toxicities; Incidence of all grades of peripheral neuropathy)

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No